CLINICAL TRIAL: NCT01993173
Title: Immunogenicity and Safety of Sanofi Pasteur's Tdap Combined Vaccine (ADACEL) as a Booster Dose, Versus Local DT Vaccine in Healthy Children or Versus Local Td Vaccine in Healthy Adolescents and Adults in China
Brief Title: Sanofi Pasteur's Tdap Combined Vaccine as a Booster Versus Local DT Vaccine in Children or Versus Local Td Vaccine in Adolescents and Adults in China.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Td528; U1111-1127-7835 (Other: WHO)
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Diphtheria; Tetanus; Pertussis
Keywords: Diphtheria; Tetanus; Pertussis; ADACEL®; Tdap vaccine
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough | interventions — Tetanus Toxoid; adacel; Diphtheria-Tetanus Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADACEL Vaccine Group (Experimental): Children, adolescents and adults randomized to receive a single booster dose of ADACEL (Tdap vaccine)
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Tdap (ADACEL)
- Local DT/Td Vaccine Group (Active Comparator): Participants randomized to receive either a single booster dose of local DT vaccine (children aged 4 through 11 years) or local Td vaccine (adolescents and adults aged 12 through 64 years)
  Interventions: Biological: DT vaccine (Diphtheria and Tetanus Combined Vaccine, Adsorbed); Biological: Td vaccine (Diphtheria and Tetanus Combined Vaccine for Adults and Adolescents, Adsorbed)

INTERVENTIONS:
Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Tdap (ADACEL) — 0.5 mL, Intramuscular
  Other Names: ADACEL
  Arms: ADACEL Vaccine Group
Biological: DT vaccine (Diphtheria and Tetanus Combined Vaccine, Adsorbed) — 0.5 mL, Intramuscular
  Arms: Local DT/Td Vaccine Group
Biological: Td vaccine (Diphtheria and Tetanus Combined Vaccine for Adults and Adolescents, Adsorbed) — 0.5 mL, Intramuscular
  Arms: Local DT/Td Vaccine Group

SUMMARY:
The aim of the study is to assess the immunogenicity and safety profile of ADACEL compared to local adsorbed diphtheria and tetanus combined vaccine (local DT or local Td vaccine in participants in China.

Primary objective:

* To describe diphtheria and tetanus seroprotection rates and pertussis booster response rates induced by each of the study vaccines: ADACEL vaccine (in all study age groups), local DT vaccine (in children), and local Td vaccine (in adolescents and adults).

Secondary Objectives:

* To further describe in each group the immunogenicity of the study vaccines at baseline and 1 month after vaccination.
* To describe the safety of the study vaccines

DETAILED DESCRIPTION:
Study participants will receive a single booster dose of ADACEL (Tdap vaccine) or a single booster dose of local DT or local Td vaccine, depending on the age subgroup.

Immunogenicity will be assessed before and 28 days post-vaccination; safety profile will be assessed in all subjects up to Day 35 post vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 4 through 64 years on day of inclusion
* For children and adolescents (4 through 17 years): Informed consent form has been signed and dated by the parent(s) or another legally acceptable representative and assent form has been signed and dated by the subject if aged 8 through 17 years

For adults (18 years and over): Informed consent form has been signed and dated by the subject

* Subject and parent / legally acceptable representative (for subjects up to 17 years) are able to attend all schedule visits and to comply with all trial procedures
* According to China National Immunization Recommendations, written documentation of complete primary series and fourth dose of diphtheria, tetanus, pertussis (DTP) vaccine for subjects aged 4 through 7 years and a written documentation or oral confirmation of complete primary series and fourth dose of DTP vaccine for subjects aged 8 through 64 years

Exclusion Criteria:

* Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine in the 4 weeks following the trial vaccination.
* Previous vaccination against diphtheria and tetanus disease with either the trial vaccine or another vaccine (except Tetanus-prone wound management for adults) in the past 12 months.
* Previous fifth vaccination against pertussis disease.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy.
* Known (laboratory-confirmed / self-reported) Human Immunodeficiency Virus (HIV) or Hepatitis C seropositivity.
* History of diphtheria, tetanus, or pertussis infection (confirmed either clinically, serologically or microbiologically).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* Laboratory-confirmed / self-reported thrombocytopenia, contraindicating intramuscular vaccination.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 37.1°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided.
* History of contra-indication to vaccination with pertussis containing vaccine, including:

  * Encephalopathy (e.g, coma, decreased level of consciousness, prolonged seizures) within 7 days of a previous dose of a pertussis containing vaccine that is not attributable to another identifiable cause
  * Progressive neurologic disorder, including infantile spasms, uncontrolled epilepsy, progressive encephalopathy
  * Axillary temperature >39.4°C within 48 hours not attributable to another identifiable cause
  * Collapse or shock-like state (hypotonic-hyporesponsive episode) within 48 hours.
* Prior personal history of Guillain-Barré syndrome.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.
* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the vaccination and until at least 4 weeks after the vaccination.

Ages: 4 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1440 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with anti-diphtheria antibody concentrations ≥ 0.1 international unit (IU)/mL | 28 Days post-vaccination
  Anti-diphtheria antibody concentrations will be determined by enzyme-linked immunosorbent assay (ELISA)
Percentage of participants with anti-tetanus antibody concentrations ≥ 0.1 IU/mL | 28 Days post-vaccination
  Anti-tetanus antibody concentrations will be determined by enzyme-linked immunosorbent assay (ELISA)
Percentage of participants with a booster response for antibodies to Pertussis Toxoid (PT), Filamentous hemagglutinin (FHA), pertactin (PRN), Fimbriae types 2 and 3 (FIM) following vaccination with ADACEL or Local DT or Local Td Vaccine | Day 0 (pre-vaccination) and Day 28 post-vaccination
  Booster response for antibodies to Pertussis Toxoid (PT), Filamentous hemagglutinin (FHA), pertactin (PRN), Fimbriae types 2 and 3 (FIM) will be determined by enzyme-linked immunosorbent assay (ELISA)

SECONDARY OUTCOMES:
Percentage of participants with anti diphtheria antibody concentrations ≥ 0.1 international unit (IU)/mL at baseline | Day 0 (pre-vaccination)
  Anti-diphtheria antibody concentrations will be determined by enzyme-linked immunosorbent assay (ELISA)
Percentage of participants with anti-tetanus antibody concentrations ≥ 0.1 IU/mL at baseline | Day 0 (pre-vaccination)
  Anti-tetanus antibody concentrations will be determined by enzyme-linked immunosorbent assay (ELISA)
Percentage of participants with anti-diphtheria antibody concentrations ≥ 1.0 international unit (IU)/mL at baseline and post booster vaccination | Day 0 (pre-vaccination) and Day 28 post-vaccination
  Anti-diphtheria antibody concentrations will be determined by enzyme-linked immunosorbent assay (ELISA)
Percentage of participants with anti-tetanus antibody concentrations ≥ 1.0 IU/mL at baseline and post booster vaccination | Day 0 (pre-vaccination) and Day 28 post-vaccination
  Anti-tetanus antibody concentrations will be determined by enzyme-linked immunosorbent assay (ELISA)
Geometric mean of individual antibody concentrations at baseline and post-booster vaccination | Day 0 (pre-vaccination) and Day 28 post-vaccination
  Antibody concentrations to all vaccine antigens will be determined by enzyme-linked immunosorbent assay (ELISA)
Number of participants reporting solicited injection site reactions, solicited systemic reactions, unsolicited adverse reactions, and serious adverse events occurring during the trial | Day 0 up to Day 28 post-vaccination
  Solicited injection site reactions: Pain, Erythema, and Swelling. Solicited systemic reactions: Fever (temperature), Headache, Malaise, and Myalgia

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Yandu, China

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com